CLINICAL TRIAL: NCT01695746
Title: Efficacy of Methoxy Poly-Ethylene Glycol Epoetin Beta (C.E.R.A.) for Correction of Anemia and Maintenance of the Hb Levels in CKD Patients in Stage III - IV, Not on Dialysis, Treated According to Routine Clinical Practice
Brief Title: An Observational Study of Mircera (Methoxy Polyethylene Glycol-Epoetin Beta) in Stage III-IV Chronic Kidney Disease Patients Not on Dialysis With Renal Anemia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25476
Record Dates: First submitted 2012-09-27; First posted 2012-09-28 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- C.E.R.A.: Participants with chronic renal anemia Stage III-IV, not on dialysis, will be administered Continuous Erythropoietin Receptor Activator (C.E.R.A.) according to routine clinical practice and will be followed up for the treatment duration of 24 weeks (6 months). Dosing and titration of C.E.R.A. treatment will be at the discretion of the investigator in accordance with local clinical practice or prescribing information. Dosing instructions as per the local label are - For correction of anemia: 0.6 microgram per kilogram (mcg/kg) of C.E.R.A. once every two weeks, and for Maintenance of hemoglobin (Hb) levels: Conversion to C.E.R.A. dose (120, 200, or 360 mcg either once monthly; or 60, 100, or 180 mcg once every 2 weeks) depending on the previous weekly epoetin or darbepoetin dose.
  Interventions: Drug: C.E.R.A.

INTERVENTIONS:
Drug: C.E.R.A. — Participants receiving 0.6 mcg/kg of C.E.R.A. once every two weeks for correction of anemia and conversion to C.E.R.A. dose 120, 200, or 360 mcg either once monthly; or 60, 100, or 180 mcg once every 2 weeks for maintenance of Hb according to local clinical practice or prescribing information will be observed.

SUMMARY:
This observational study will evaluate the use in clinical practice and efficacy of Mircera (methoxy polyethylene glycol-epoetin beta) in stage III-IV chronic kidney disease patients not on dialysis receiving Mircera for the treatment of chronic renal anemia. Eligible patients will be followed for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 65 years of age, inclusive
* Patients with stage III-IV chronic kidney disease not on dialysis
* Erythropoiesis stimulating agent (ESA) naïve with Hb < 10 g/dL, or on treatment with ESAs other than Mircera and Hb within the target range of 10-12 g/dL
* Adequate iron status as judged by the treating physician

Exclusion Criteria:

* Hypersensitivity to recombinant human erythropoietin, polyethylene glycol or to any constituent of the study medication
* Clinically significant concomitant disease or disorder as defined by protocol
* Clinical suspicion of pure red cell aplasia (PRCA)
* Planned elective surgery during the study period , except for cataract surgery or vascular access surgery
* Transfusion of red blood cells in the previous 2 months
* Pregnant women
* Contraindications for Mircera according to local prescribing information or as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage III-IV chronic kidney disease not on dialysis receiving treatment with Mircera for chronic renal anemia
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- India (5):
  - Bhubaneswar
  - Hyderabad
  - Mumbai
  - Vadodara
  - Vellore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 108 participants were enrolled in this study conducted from 30 August 2011 to 13 November 2013 at 6 sites in India.
Groups:
- C.E.R.A.: Participants with chronic renal anemia Stage III-IV, not on dialysis, were administered C.E.R.A. according to routine clinical practice and were followed for the treatment duration of 24 weeks (6 months). Dosing and titration of C.E.R.A. treatment was at the discretion of the investigator in accordance with local clinical practice or prescribing information. Dosing instructions as per the local label were - For correction of anemia: 0.6 mcg/kg of C.E.R.A. once every two weeks, and for Maintenance of Hb levels: Conversion to C.E.R.A. dose (120, 200, or 360 mcg either once monthly; or 60, 100, or 180 mcg once every 2 weeks) depending on the previous weekly epoetin or darbepoetin dose.
Period: Overall Study
Arm/Group | C.E.R.A.
Started | 108
Completed | 96
Not Completed | 12
Not completed — Adverse Event | 1
Not completed — Non-compliance by the participant | 3
Not completed — Protocol Violation | 5
Not completed — Participant not willing to participate | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were evaluated for the safety population which included all participants entered into the study.
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (7.178)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 72

OUTCOME MEASURES:

1. Primary Outcome: Mean Height of Participants at Baseline (Week 0)
Description: The mean body height of the participants was measured and summarized in centimeters (cm). Baseline is defined as Week 0.
Time Frame: At Baseline (Week 0)
Population: The safety population included all participants entered into the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 108
cm | 163.15 (7.366)

2. Primary Outcome: Mean Weight of Participants at Baseline (Week 0)
Description: The mean body weight of the participants was measured and summarized in kg. Baseline is defined as Week 0.
Time Frame: At Baseline (Week 0)
Population: The safety population included all participants entered into the study.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 108
kg | 60.23 (9.618)

3. Secondary Outcome: Percentage of Participants Achieving Hemoglobin Target Range (10-12 Gram/Deciliter) at Least Once During the Study
Description: Correction of anemia was evaluated in participants with Hb < 10 g/dL at enrollment. Hemoglobin levels were recorded for each participant at enrollment and at different time points during the study up to Week 24. The percentage of participants achieving the target Hb range (10-12 g/dL) at least once during the study is presented.
Time Frame: Up to Week 24
Population: The ITT population included all participants who received at least 1 dose of C.E.R.A. (Week 0), for whom data for at least one follow-up variable was available, and who did not have a major protocol violation.
Measure: Number; unit: Percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 92
Percentage of participants | 90.2

4. Secondary Outcome: Mean Time Spent in the Hemoglobin Target Range (10 - 12 Gram/Deciliter)
Description: The Hb concentration was recorded for all the participants at enrollment and different time points throughout the study up to Week 24. The mean time spent (in weeks) by the participants in the target range (10 - 12 g/dL) is presented.
Time Frame: Up to Week 24
Population: The ITT population included all participants who received at least 1 dose of C.E.R.A. (Week 0), for whom data for at least one follow-up variable was available, and who did not have a major protocol violation. The participants who achieved target Hb range (10-12 g/dL) were included in the analysis.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 72
Weeks | 16.69 (4.124)

5. Secondary Outcome: Mean Dose of C.E.R.A. Administered
Description: The mean dose of C.E.R.A. administered during the study is reported. This accounts for the study drug injected through subcutaneous route at a frequency of every 4 weeks or once a month and every 2 weeks or fortnightly.
Time Frame: Up to Week 24
Population: The safety population included all participants entered into the study.
Measure: Mean (Standard Deviation); unit: mcg per month
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 108
mcg per month | 75.5 (26.79)

6. Secondary Outcome: Number of Doses of C.E.R.A. Administered by Different Routes
Description: The number of doses of C.E.R.A. administered by the intravenous or subcutaneous route is presented. The number of doses for total population is calculated by summation and presented in table below as per routes of administration.
Time Frame: Up to Week 24
Population: The safety population included all participants entered into the study.
Measure: Number; unit: Doses
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 108
Doses
  Intravenous route | 0
  Subcutaneous route | 572

7. Primary Outcome: Number of Participants With Co-morbidities at Baseline (Week 0)
Description: Co-morbidities were those medical disorders present in the medical history but unresolved at Baseline. The number of participants with different co-morbidities is presented. Baseline is defined as Week 0.
Time Frame: At Baseline (Week 0)
Population: The safety population included all participants entered into the study.
Measure: Number; unit: Participants
Groups:
- C.E.R.A (Continuous Erythropoietin Receptor Activator): Participants with chronic renal anemia Stage III-IV, not on dialysis, receiving therapy with C.E.R.A. according to routine clinical practice were followed for the treatment duration of 24 weeks (6 months). Dosing and titration of C.E.R.A. treatment was at the discretion of the investigator in accordance with local clinical practice or prescribing information. Dosing instructions as per the local label were - For correction of anemia: 0.6 μg/kg of C.E.R.A once every two weeks, and for Maintenance of Hb levels: Conversion to C.E.R.A. dose (120, 200, or 360 μg either once monthly; or 60, 100, or 180 μg once every 2 weeks) depending on the previous weekly epoetin or darbepoetin dose.
Arm/Group | C.E.R.A (Continuous Erythropoietin Receptor Activator)
Number analyzed (Participants) | 108
Participants
  Anaemia | 2
  Myocardial ischaemia | 4
  Congenital cystic kidney disease | 1
  Renal hypoplasia | 1
  Hypothyroidism | 4
  Liver disorder | 1
  Diabetes mellitus | 18
  Dyslipidaemia | 1
  Type 1 diabetes mellitus | 1
  Type 2 diabetes mellitus | 66
  Osteoarthritis | 2
  Osteoporosis | 1
  Rheumatoid arthritis | 1
  Systemic lupus erythematosus | 1
  Glomerulonephritis | 2
  Nephrolithiasis | 2
  Nephropathy | 1
  Renal failure chronic | 28
  Tubulointerstitial nephritis | 1
  Asthma | 1
  Chronic obstructive pulmonary disorders | 1
  Coronary angioplasty | 1
  Renal transplant | 1
  Hypertension | 90

8. Primary Outcome: Mean Time to Achieve Target Hemoglobin Range (10-12 Gram/Deciliter)
Description: Correction of anemia was evaluated in participants with Hb < 10 gram/deciliter (g/dL). Hemoglobin levels were recorded for each participant at enrollment and at different time points during the study up to Week 24. The mean time required to achieve target Hb range (10-12 g/dL) was calculated using the following formula: Time to achieve target range = (Date of Hb evaluation when participant achieves target range at first time - visit date of first dosing) + 1.
Time Frame: Up to Week 24
Population: The intent-to-treat (ITT) population included all participants who received at least 1 dose of C.E.R.A. (Week 0), for whom data for at least one follow-up variable was available, and who did not have a major protocol violation. The participants who achieved target Hb range (10-12 g/dL) were included in the analysis.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 83
Weeks | 9.61 (6.130)

9. Primary Outcome: Percentage of Participants Maintaining Hemoglobin Level Within 1 Gram/Deciliter of Baseline Value
Description: Maintenance of Hb levels was to be evaluated for participants on Erythropoiesis stimulating agent (ESA) with Hb levels 10-12 g/dL. None of the participants in the enrolled population had received treatment with other ESAs and had pre-therapy Hb level as 10 g/dL or above. Therefore, the percentage of participants who had received treatment with other ESAs and were maintaining Hb level within 1 g/dL of baseline value during the study could not be evaluated. Baseline is defined as Week 0.
Time Frame: Up to Week 24
Population: The ITT population was the anticipated population for analysis.
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Participants Who Received Concomitant Treatment for Anemia
Description: Medications that were used during the study treatment period (from the date of first dose of study medication to the end of the study) were included as concomitant medications. The number of participants taking concomitant medications prescribed for the treatment of anemia (for example iron) is presented.
Time Frame: Up to Week 24
Population: The safety population included all participants entered into the study.
Measure: Number; unit: Participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 108
Participants
  Multivitamin | 17
  Iron supplement | 15
  Vitamin B | 15
  Iron + multivitamin | 2

11. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Pre-existing conditions which worsened during this study were reported as AEs. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Week 24
Population: The safety population was defined as all participants entered into the study.
Measure: Number; unit: Participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 108
Participants
  Number of participants with any AE | 4
  Number of participants with any SAE | 2

ADVERSE EVENTS:
Time Frame: Up to Week 24
Description: Adverse event data was reported for the safety population which included all participants entered into the study.
Arm/Group | C.E.R.A.
Serious Adverse Events (participants affected / at risk) | 2/108
Other Adverse Events (participants affected / at risk) | 2/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=108)
Pancreatitis (Gastrointestinal disorders) | 1
Device related infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=108)
Nasopharyngitis (Infections and infestations) | 1
HIV test positive (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.